CLINICAL TRIAL: NCT02435979
Title: Proximal Strengthening for the Management of Wrist Pain: A Randomized Controlled Trial
Brief Title: Proximal Strengthening for the Management of Wrist Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitchell Selhorst (Other)
Responsible Party: Sponsor-Investigator, Mitchell Selhorst, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-00251
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Wrist Injuries
Keywords: wrist; proximal strengthening; hand therapy
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proximal strengthening + hand therapy (Experimental): Patients in this group will perform traditional hand therapy for 30 minutes and proximal strengthening of the core, cervical spine, and shoulder complex for up to 30 minutes
  Interventions: Other: hand therapy; Other: Proximal Strengthening
- Traditional hand therapy (Active Comparator): This group will receive traditional hand therapy for 45-60 minutes each session.
  Interventions: Other: hand therapy

INTERVENTIONS:
Other: hand therapy — Treatment can include stretching, motion, and strengthening exercises. As the patients endurance and strength increased the repetitions and/or resistance of these exercises will increase. Modalities for pain control and tissue mobility, and bracing or splinting if necessary. All treatments for the traditional hand therapy treatment group will occur seated at the hand therapy treatment table.
Other: Proximal Strengthening — Patients will perform a standardized proximal strengthening protocol consisting of cervical, periscapular, and shoulder strengthening exercises. Depending on the pace and guidance needed for these exercises 25-30 minutes will be spent on proximal strengthening exercises. As the patients endurance and strength increased the repetitions and/or resistance of these exercises will increase.
  Arms: Proximal strengthening + hand therapy

SUMMARY:
This study will be a randomized controlled trial comparing proximal strengthening vs. traditional hand therapy for patients with wrist pain. Patients will attend 2 hand therapy sessions per week for 4 weeks. Change in patient function and pain as measured by the patient rated wrist evaluation will be the primary outcome of interest

DETAILED DESCRIPTION:
This will be a non-blinded randomized controlled trial using a sample of consecutive patients with wrist pain. Patients who are referred to Nationwide Children's Hospital Hand therapy clinics with a primary complaint of wrist pain will be considered for this study.

Patients will be randomly assigned to one of two treatment groups; The proximal strengthening group or Traditional Hand Therapy Group. Both treatment groups will be evaluated and treated by the certified hand therapists for 2 sessions per week for 4 weeks. Both groups will receive similar treatment durations of 45-60 minutes per session based on each patient's individual needs.

Proximal strengthening group-The experimental proximal strengthening group consists of treatment where the hand therapist address specific impairments at the wrist and hand for 20-30 minutes at each treatment session. Patients allocated to this treatment group will also perform a standardized proximal strengthening protocol consisting of cervical, periscapular, and shoulder strengthening exercises. Depending on the pace and guidance needed for these exercises 25-30 minutes will be spent on proximal strengthening exercises. As the patients endurance and strength increased the repetitions and/or resistance of these exercises will increase.

Traditional Hand Therapy Group This active comparator group consists of treatment where the hand therapist address specific impairments at the wrist and hand for 45-60 minutes at each treatment session. Treatment can include stretching, motion, and strengthening exercises. As the patients endurance and strength increased the repetitions and/or resistance of these exercises will increase. Modalities for pain control and tissue mobility, and bracing or splinting if necessary. All treatments for the traditional hand therapy treatment group will occur seated at the hand therapy treatment table.

ELIGIBILITY:
Inclusion Criteria:

* Wrist pain

Exclusion Criteria:

* <8 years of age
* any neurological disorder
* Juvenile rheumatoid arthritis
* juvenile idiopathic arthritis
* Wrist fractures < 16 weeks from date of injury or surgery
* Tendon repair
* Nerve injury or repair
* Inability to follow directions
* Inability to attend follow-up appointments

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in Patient Rated Wrist Evaluation (PRWE) score | 4 weeks (From initial evaluation to discharge)
  The PRWE is a 15 item self-report questionnaire which measure pain and function. It has been found valid and reliable for measure changes in pain and function for patients with wrist pain. The minimal clinical important difference of this scale is 14 (Sorensen, 2013).

SECONDARY OUTCOMES:
Change in Grip Dynamometer strength | 4 weeks (From initial evaluation to discharge)
  Grip strength will be measured using a Jamar dynamometer on 2nd setting with elbow at 90 deg and shoulder in adduction at the patient's side, with the patient seated. Grip strength will be expressed as a percentage of body weight to account for differences in patients size and strength.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Childrens Hospital
Locations (4):
- United States (4):
  - Nationwide Children's Hospital Sports and Ortho PT Ortho Center, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Dublin, Dublin, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio

REFERENCES:
- [Background] Alexander M, Franko OI, Makhni EC, Zurakowski D, Day CS. Validation of a modern activity hand survey with respect to reliability, construct and criterion validity. J Hand Surg Eur Vol. 2008 Oct;33(5):653-60. doi: 10.1177/1753193408093810. PMID 18977836
- [Background] Metzler W, Kessler G, Benzer W, Mahr G. [Ophthalmological significance of stenosing carotid processes]. Wien Med Wochenschr. 1990 Jul 31;140(14):387-9. German. PMID 2219945
- [Background] Emery K, De Serres SJ, McMillan A, Cote JN. The effects of a Pilates training program on arm-trunk posture and movement. Clin Biomech (Bristol). 2010 Feb;25(2):124-30. doi: 10.1016/j.clinbiomech.2009.10.003. Epub 2009 Oct 30. PMID 19879677
- [Background] Kalra N, Seitz AL, Boardman ND 3rd, Michener LA. Effect of posture on acromiohumeral distance with arm elevation in subjects with and without rotator cuff disease using ultrasonography. J Orthop Sports Phys Ther. 2010 Oct;40(10):633-40. doi: 10.2519/jospt.2010.3155. PMID 20710092
- [Background] Kong YK. The effects of co-ordinating postures with shoulder and elbow flexion angles on maximum grip strength and upper-limb muscle activity in standing and sitting postures. Int J Occup Saf Ergon. 2014;20(4):595-606. doi: 10.1080/10803548.2014.11077077. PMID 25513795
- [Background] MacDermid JC. Development of a scale for patient rating of wrist pain and disability. J Hand Ther. 1996 Apr-Jun;9(2):178-83. doi: 10.1016/s0894-1130(96)80076-7. No abstract available. PMID 8784681
- [Background] Park JK, Buchholz B. Effects of work surface height on muscle activity and posture of the upper extremity during simulated pipetting. Ergonomics. 2013;56(7):1147-58. doi: 10.1080/00140139.2013.799234. Epub 2013 Jun 6. PMID 23742175
- [Result] Sorensen AA, Howard D, Tan WH, Ketchersid J, Calfee RP. Minimal clinically important differences of 3 patient-rated outcomes instruments. J Hand Surg Am. 2013 Apr;38(4):641-9. doi: 10.1016/j.jhsa.2012.12.032. Epub 2013 Mar 6. PMID 23481405